CLINICAL TRIAL: NCT00167115
Title: Metabolic Effects of Alcohol in the Form of Wine in Persons With Type 2 Diabetes Mellitus
Brief Title: Metabolic Effects of Alcohol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bantle, John P., MD (Individual)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0406M61001; Bantle1
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Alcohol; Type 2 diabetes mellitus; Plama glucose; HDL cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alcohol

SUMMARY:
The hypotheses to be tested are 1) the use of alcohol in the form of wine with the evening meal will lower plasma glucose during the night and result in lower fasting plasma glucose the next morning; 2) the chronic use of alcohol in moderation in the form of wine will have beneficial effects on plasma lipids in type 2 diabetic subjects.

DETAILED DESCRIPTION:
The use of alcohol in moderation has been associated with reduced mortality rates, reduced risk of cardiovascular disease and reduced risk for type 2 diabetes. However, the effects of alcohol in persons with type 2 diabetes have not yet been defined. Moreover, the possibility of alcohol induced hypoglycemia remains a safety concern. Finally, little is known about the effects of alcohol on plasma lipids in people with diabetes. To address these issues, two substudies are proposed. The first substudy will examine the acute effects of alcohol in the form of wine at supper on postprandial and nocturnal glucose levels. The second substudy will examine the effects of alcohol in the form of wine consumed regularly for one month on plasma lipids.

To test these hypotheses, 20 type 2 diabetics will be studied. In substudy 1, subjects will be admitted to the Clinical Research Center for a two day inpatient stay. Blood samples for plasma glucose and serum insulin will be obtained every two hours from 5:00 pm to 7:00 am. On one day, subjects will recieve 8 ounces of wine with dinner. On the other day, subjects will recieve 8 ounces of fruit juice with dinner. The primary endpoint of substudy 1 will be fasting plasma glucose. In substudy 2, subjects will be asked to consume 4-8 ounces of wine in the evening for one month and to abstain from wine and alcohol containing beverages for one month. Fasting blood samples will be obtained after the month of wine consumption and after the month of abstention from alcohol for measurement of fasting lipids. The primary endpoint of substudy 2 will be fasting HDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes HbA1c 6.0-8.0% age > 40 years

Exclusion Criteria:

History of alcoholism or alcohol abuse liver disease blood pressure > 150/90

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Fasing plasma glucose
Fasting plasma HDL cholesterol

SECONDARY OUTCOMES:
Episodes of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: John Bantle, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States